CLINICAL TRIAL: NCT06783179
Title: Postoperative Outcomes and Patient Satisfaction for Patients Admitted to the Mayo Clinic Florida Care Hotel After Mastectomy and Tissue Expander Placement
Brief Title: Postoperative Outcomes and Patient Satisfaction With Mayo Clinic Florida Care Hotel After Mastectomy and Tissue Expander Placement
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 24-006876; NCI-2024-10631 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-006876 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients have their medical records reviewed and may complete a survey on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates the postoperative outcomes of patients who are admitted to the Mayo Clinic Florida Care Hotel after mastectomy and tissue expander placement. At Mayo Clinic Florida, patients receiving low risk surgeries are often admitted to the hospital overnight for observation. A new model of delivering patient care was created at the Mayo Clinic Florida coined the "Care Hotel." This is a temporal, voluntary accommodation that offers patients a comfortable environment to receive nursing care before or after hospital treatment with in-person daytime monitoring and 24-hour virtual tele-monitoring in a hotel setting. This study evaluates post operative complications in patients who underwent mastectomy followed by tissue expander reconstruction and were admitted to the Care Hotel for overnight observation compared to the standard hospital admission and those who are discharged home.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate post operative complications in patients who underwent mastectomy followed by tissue expander reconstruction and were admitted to the Care Hotel for overnight observation compared to the standard hospital admission and those who are discharged home.

OUTLINE: This is an observational study.

Patients have their medical records reviewed and may complete a survey on study.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent mastectomy followed by tissue expander reconstruction for breast cancer or high-risk gene mutation prophylaxis followed by immediate tissue expander reconstruction who are either admitted to the Care Hotel post operatively, discharge home or admitted to the hospital.

Exclusion Criteria:

* Younger than 18 years old.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who underwent mastectomy followed by tissue expander reconstruction for breast cancer or high-risk gene mutation prophylaxis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2027-12-16 (Estimated); Study Completion 2027-12-16 (Estimated)

PRIMARY OUTCOMES:
Complications | Up to 30 days
  Recorded as incidence of hematoma, infection, readmission, and/or reoperation within 30 days of initial procedure.

SECONDARY OUTCOMES:
Patient satisfaction | Up to 30 days
  Assessed via voluntary survey given at first routine post operative visit to all patients who were admitted to the Care Hotel. The survey consists of 5 questions related to the Care Hotel Stay and one question related to pain level during the stay.. The 5 questions are answered on a scale ranging from 1-5 where 1=strongly disagree and 5=strongly agree, and the final questions is answered on a scale of 1-10 where 1=little pain and 10=worst pain ever experienced. There are also free-text sections for participants to indicate anything that impressed them about their experience with Care Hotel and/or anytihng that disappointed them about their experience.

CONTACTS AND LOCATIONS:
Overall Officials: Brian D. Rinker, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials